CLINICAL TRIAL: NCT02906475
Title: A Randomized Pragmatic Parallel Group Trial to Investigate the Effectiveness of a Standardized Skin Care Regimen to Prevent the Development of Atopic Dermatitis in Atopy Predisposed Infants
Brief Title: Atopic Dermatitis in Atopy Predisposed Infants
Acronym: ADAPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HiPP GmbH & Co. Vertrieb KG (Industry)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 508276
Record Dates: First submitted 2016-09-15; First posted 2016-09-20 (Estimated); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Dermatitis, Atopic
Keywords: Dermatitis, atopic; prevention and control; Infant; Skin care; randomized controlled trial
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention: standardized skin care regimen (Other): Intervention: The milk lotion will be applied once daily on the total body including the face by the parents or care givers at home. If bathing is needed, the bathing addendum is used in addition to water.
  Interventions: Other: standardized skin care regimen
- Control (No Intervention): In the control group no predetermined or standardized skin care regimen is prescribed.

INTERVENTIONS:
Other: standardized skin care regimen — Application of a standardized daily skin care regimen:
  * milk lotion once daily and
  * application of addendum for bathing as needed
  Arms: Intervention: standardized skin care regimen

SUMMARY:
The primary objective of this study is to investigate the effectiveness of a standardized skin care regimen using a milk lotion once daily and a bathing addendum as needed during the first 52 weeks of life on the development of atopic Dermatitis (AD) compared to no structured skin care regimen in infants with atopic predisposition. Secondary objectives are to investigate the influence of a structured skin care regimen on the development of AD in the second year of life and the skin barrier function up to the infants' age of 2 years.

DETAILED DESCRIPTION:
Atopic dermatitis is the most common cutaneous disease in childhood. First manifestations of AD usually appear early in life after the 3rd month of life and often precede other allergic diseases such as asthma or allergic rhinitis. AD affects over 15% of children up to school age in Germany and has a substantial impact on the lives and life quality of both the child and its family. Taking into account the burden on health-care resources, the impact on the quality of life of patients and their caregivers, together with increasing evidence that AD may progress to other allergic phenotypes, there is a clear need to improve disease prevention. Due to the childhood prevalence of the disease, prevention is focused on the postnatal period. It is recognized that prevention should start as soon as possible. Current studies suggest that epidermal barrier impairment is an important factor for the development of AD and other allergic diseases, with the gene encoding the filament-binding protein filaggrin (FLG) being the most widely replicated and most significant gene to influence atopic diseases. Currently, no standardized recommendations for preventive therapies exist for AD. Pilot studies have focused on interventions to enhance skin barrier function. Daily skin care with an emollient early after birth is considered to reduce the risk of atopic dermatitis in infants.

The study will be divided in 2 parts: The main study (Interventional period) lasts up to the child´s age of one year (52 weeks of life) and the follow-up period up to the second birthday.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent (by both parents or legal representatives)
2. Healthy term newborns (gestational age: completed 37 weeks) born by mothers aged 18-45 years
3. Birth weight between 2.500 - 4.500 g
4. Age at enrolment 14 days
5. Infants at enhanced risk for developing AD (at least one parent or sibling with physician-diagnosed AD, asthma or allergic rhinitis/rhino conjunctivitis as reported by at least by one parent but in otherwise good overall health
6. Infant Nutrition: breastfeeding or cow's-milk based infant formula (including Hypoallergenic (HA) - based formula) feeding or combination
7. Phototype I, II, III or IV according to the Fitzpatrick classification.

Exclusion Criteria:

1. Serious acquired or congenital diseases
2. Hydrops fetalis
3. Preterm children (< completed 37th week of gestation)
4. Weight at birth < 2500 g or > 4500 g
5. Significant dermatitis at birth except seborrheic dermatitis on the scalp ("cradle cap")
6. Dermatological conditions influencing the study parameters, besides benign transient neonatal diseases
7. Any immunodeficiency disorder
8. Any severe genetic skin disorder
9. Any other serious condition that would make the use of skin care products inadvisable
10. Any other major medical problems that the investigator deems may increase the risk of adverse events with the intervention or in whom assessing the outcomes may be masked by the underlying problem or practically very difficult to assess
11. Participation in another clinical study
12. Reason to presume that the parents are unable to meet the study plan requirements
13. Nutrition: other than breastfeeding or cow's-milk based infant formula (e.g. soybased, goat-milk based formula etc.)
14. History of allergy or intolerance to investigational product's ingredient(s) of at least one subject's parent
15. Current topical or systemic drug treatment
16. Maternal antibiotic therapy in breastfed newborns
17. Infants of mothers supplementing probiotics during pregnancy and/or breastfeeding on a regular basis

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of atopic dermatitis | 12 months
  Cumulative incidence of AD at week 52, with AD diagnosis based on the criteria by Simpson et al. 2012

SECONDARY OUTCOMES:
Cumulative incidence of atopic dermatitis | 24 months
AD incidence density | 12 months
AD incidence density | 24 months
Eczema Area and Severity Index (EASI) | 12 months
Eczema Area and Severity Index (EASI) | 24 months
Infant Dermatitis Quality of Life (IDQoL) | 12 months
Infant Dermatitis Quality of Life (IDQoL) | 24 months
Transepidermal water loss (TEWL) on the midvolar forearm | at ages of 14 days, 1, 3, 6, 12 months and 2 years
Skin surface pH on the midvolar forearm | at ages of 14 days, 1, 3, 6, 12 months and 2 years
Stratum Corneum Hydration (SCH) on the forearm | at ages of 14 days, 1, 3, 6, 12 months and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Blume-Peytavi, Prof. Dr., Principal Investigator — Charite Universitätsmedizin Berlin
Locations (1):
- Charite Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simpson EL, Keck LE, Chalmers JR, Williams HC. How should an incident case of atopic dermatitis be defined? A systematic review of primary prevention studies. J Allergy Clin Immunol. 2012 Jul;130(1):137-44. doi: 10.1016/j.jaci.2012.01.075. Epub 2012 Mar 15. PMID 22424882